CLINICAL TRIAL: NCT05116254
Title: Sarcomas and DDR-Inhibition; a Neoadjuvant Phase I Combined Modality Study.
Brief Title: Sarcomas and DDR-Inhibition; a Combined Modality Study
Acronym: SADDRIN-1
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Endpoint has been reached.
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Leiden University Medical Center (Other); University Medical Center Nijmegen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M21SAD
Record Dates: First submitted 2021-10-14; First posted 2021-11-10 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Soft Tissue Sarcoma Adult
Keywords: soft tissue sarcoma; radiotherapy; DNA Damage Response
MeSH Terms: conditions — Sarcoma | interventions — AZD1390; Radiotherapy

STUDY DESIGN:
Intervention Model Description: I: AZD1390 and RT II: AZD1390, durvalumab and RT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AZD1390 (Other): The experimental oral drug AZD1390 (starting dose once daily 20 mg) will be combined with radiotherapy. Drug will be taken at same day as radiotherapy for 5 weeks at weekdays.
  When starting dose of 20 mg is proven safe the next cohort will be 100 and thereafter 200, 400 mg
  Interventions: Combination Product: AZD1390 + radiotherapy
- AZD1390 + durvalumab (Other): The experimental oral drug AZD1390 (starting dose once daily 20 mg) will be combined with radiotherapy and durvalumab (fixed dose 1500 mg Q4W, until surgery). Drug will be taken at same day as radiotherapy for 5 weeks at weekdays. The dose of AZD1390 in the AZD1390 plus durvalumab cohort will follow the dosing of the AZD1390 only cohort. When starting dose of 20 mg and the next dose of AZD1390 only has been proven safe, the next cohort will be 100 and thereafter 200, 400 mg.
  Interventions: Combination Product: AZD1390 + durvlaumab + radiotherapy

INTERVENTIONS:
Combination Product: AZD1390 + radiotherapy — AZD1390 combined with preoperative radiotherapy
  Arms: AZD1390
Combination Product: AZD1390 + durvlaumab + radiotherapy — AZD1390 combined with durvalumab and preoperative radiotherapy
  Arms: AZD1390 + durvalumab

SUMMARY:
To assess the safety and tolerability profile, in the pre- and perioperative period (up to 30 days post-surgery), of combined modality treatment (CMT) by administering AZD1390 with or without durvalumab and RT concurrently treating newly diagnosed, non-metastatic soft tissue sarcoma patients with DDRi-based CMT, in the specific context of systemic toxicities, wound healing post-surgery and in defining the RP2D for the combinations to support further clinical evaluation.

DETAILED DESCRIPTION:
Despite improvements in surgery and radiation for soft tissue sarcoma (STS) patients, local relapses remain an important event for these patients. Most STS subtypes are considered radioresistant and immune cold tumor due to a lack of T-cell infiltration. Investigations into radiosensitization mediated by combining systemic compounds with neoadjuvant radiotherapy (RT) may translate into an increased rate of pathological responses, an increased rate of R0 resections and thus fewer local relapses.

RT is highly potent in inducing DNA damage. Normal cells are usually sufficiently able to repair this damage timely before the next fraction because of an intact DNA Damage Response (DDR) pathway. Frequently, tumor cells have (partial or complete) defects in the DDR pathways rendering them more sensitive to radiation than normal tissues. Inhibition of constituents of the DDR pathways may further widen the therapeutic window of fractionated radiotherapy, and combined with radiotherapy may result in increased tumor T-cell infiltration, creating an opportunity for immunotherapy. Clinical studies into radiosensitization of STS by combinations of radiotherapy and DDR inhibitors with or without immunotherapy are warranted. In this study the DDR candidate inhibitor is new drug candidate AZD1390 targeting ATM (Ataxia Telangiectasia Mutated). The immunotherapy candidate of this study is durvalumab (MEDI4736) targeting PD-L1 (programmed death-ligand 1).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed newly diagnosed intermediate to high grade soft tissue sarcoma localized to the extremities, for which the standard treatment is a combination of RT and surgery (in other words deep seated and/or > 5cm in largest tumor diameter and/or an anticipated close resection margin and/or grade II/III according to the FNCLCC definition);
* Patients staged by at least a CT scan of the chest (and a CT scan of the abdomen, if deemed indicated according to local practices, e.g. in case of a myxoid liposarcoma). Staging may also be performed by FDG-PET scanning and or total body MRI scans. This staging procedure should not reveal metastatic disease. If, however, a low metastatic burden is detected such that this does not preclude the application of both preoperative RT and definitive surgery, patients are allowed to participate;
* WHO Performance Status ≤ 2;
* Able and willing to undergo preoperative RT;
* Able and willing to undergo definitive surgery;
* Able and willing to comply with regular follow-up visits;
* Able and willing to swallow and retain oral medication;
* Age ≥ 18 years;
* Body weight >30kg;
* Must have a life expectancy of at least 12 weeks;
* Adequate organ function as defined in Table 5;
* Signed written informed consent prior to any study specific procedures or sampling

Exclusion Criteria:

* Patients with any type soft tissue sarcoma located above the clavicles.
* Prior malignancies; except another malignancy and disease-free for ≥ 5 years, or completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma;
* Patients with recurrent sarcomas who underwent prior RT to the target lesion (if the primary sarcoma was managed by surgery only and no perioperative RT, patients are eligible);
* Ewing sarcoma and other PNET family tumors, rhabdomyosarcomas (both pediatric and adult), bone sarcomas;
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial;
* Female patients who are pregnant or breast feeding;
* Intention to perform an isolated limb perfusion, instead of a tumor resection;
* Neoadjuvant chemotherapy to be scheduled between end of RT and definitive surgery is not allowed. (neoadjuvant chemotherapy before start of study RT is allowed);
* Concomitant treatment with medicines listed as 'prohibited' or 'excluded';
* Treatment with moderate and strong inhibitors or inducers of CYP3A4 within 2 weeks before the first dose of study treatment (3 weeks for St John's Wort);

Additional criteria for durvalumab plus AZD1390:

* Past medical history of allogenic organ transplantation;
* Past medical history of leptomeningeal carcinomatosis;
* Past medical history or active autoimmune or inflammatory disorders
* History or presence of primary immunodeficiency
* Presence of active hepatitis infections or HIV
* Treatment with or prior use of immunosuppressive medication within 2 weeks before the start of treatment
* Prior treatment with anti-PD-1, anti PD-L1 or anti CTLA-4 immunotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2025-12-09 (Actual); Study Completion 2025-12-09 (Actual)

PRIMARY OUTCOMES:
Drug safety | 2 years
  all adverse events
Drug tolerability | 30 days
  adverse events and more specific woundhealing

SECONDARY OUTCOMES:
Tumor regression | After 5 weeks of RT and DDRi-based drug treatment
  pathological remission
Local control rates | 2 years
  Histopathological response and MRI
Rate of R0 resection | Directly after surgery
  Histological examination of surgical specimens
Rate of R1 resection | Directly after surgery
  Histological examination of surgical specimens

CONTACTS AND LOCATIONS:
Overall Officials: Rick Haas, MD Prof, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- Antoni van Leeuwenhoek, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No